CLINICAL TRIAL: NCT04375735
Title: Phase I/II Trial: Exogenous Surfactant Administration for Patients With COVID-19
Brief Title: London's Exogenous Surfactant Study for COVID19
Acronym: LESSCOVID
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: London Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9890
Record Dates: First submitted 2020-04-22; First posted 2020-05-05 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: ARDS, Human; COVID-19
MeSH Terms: conditions — Respiratory Distress Syndrome; COVID-19 | interventions — Surface-Active Agents

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned to either receive exogenous surfactant daily for 3 days, or receive standard treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BLES treatment (Experimental): For patients randomized to the treatment arm, exogenous BLES will be administered as soon as possible and within 48 hours of intubation. BLES will be administered daily for up to 3 doses, or until the patient is liberated from the ventilator.
  Interventions: Drug: Bovine Lipid Extract Surfactant
- Control (No Intervention): Patients will receive standard treatment and will not receive surfactant.

INTERVENTIONS:
Drug: Bovine Lipid Extract Surfactant — BLES will be administered in doses of 50mg/kg ideal bodyweight, at a concentration of 27mg/ml so a total volume of approximately 2ml/kg will be administered. The material will be instilled via the suction catheter through the ET tube so that the ventilation circuit is not broken. Half of the material will be instilled with the patient positioned on their left and right sides, with a pause to allow 5 min of MV between. The procedure will be repeated at, 24 and 48 hours while intubated, so the patient will receive up to 3 doses. To minimize aerosol generation, all patients will be paralyzed during surfactant administration and the ventilator will be paused. The proposed administration technique, surfactant concentration, volume and dosing schedule is based on previous studies, and has shown to be safe in patients with ARDS.
  Other Names: BLES; Lung Surfactant; Bovine
  Arms: BLES treatment

SUMMARY:
The research team is investigating administering exogenous surfactant in COVID-19 patients with ARDS. The overall goal is to improve the outcome (mortality) of mechanically ventilated COVID-19 patients. Although the investigators anticipate that clinical outcomes may improve in the small group of patients receiving exogenous surfactant therapy in this small, single center study, the primary goal is to first determine feasibility and safety.

DETAILED DESCRIPTION:
The most severe patients infected by the virus that causes COVID-19 develop severe respiratory failure (called ARDS) and require mechanical ventilation in the intensive care unit to help maintain oxygen delivery to the blood. Often these patients further deteriorate while on mechanical ventilation. This trial will determine the feasibility and safety of a therapy that can potentially improve lung function, reduce the need for mechanical ventilation and hopefully impact mortality.

Adult patients with COVID-19 induced respiratory failure will be randomly assigned to receive either standard treatment or standard treatment plus exogenous surfactant. If enrolled in the latter, exogenous surfactant will be instilled into the lungs within 48 hours of intubation.

The study is founded on extensive research on ARDS for over 30 years, leading to evidence suggesting that exogenous surfactant administration may be beneficial in this disease. Importantly, exogenous surfactant is already utilized all over the world to reduce mortality in preterm infants. When tested in adults with ARDS, it was shown to be well tolerated and safe. Furthermore, clinical and laboratory evidence suggests that this therapy may be most effective in patients with a direct lung infection, and when administered shortly after the patient is intubated. In this study, twenty patients who are proven COVID-19 positive and require MV due to progressive respiratory failure will be randomized to receive either 1) exogenous surfactant (BLES) as soon as possible and within 48 hours of intubation and stabilization, or 2) treatment as usual (will not be treated with surfactant). The overall goal is to improve the outcome (mortality) of mechanically ventilated COVID-19 patients. Although the investigators anticipate that clinical outcomes may improve in the small group of patients receiving exogenous surfactant therapy in this small, single center study, the primary goal is to first determine feasibility and safety. Should the investigators obtain promising results, the data obtained from this study will be used to develop a large trial to test the impact of this therapy on the clinical outcomes, including mortality, associated with COVID-19.

ELIGIBILITY:
Inclusion Criteria:

1. age over 18 years
2. definitive proof of COVID-19 infection within 48 hours of intubation
3. acute respiratory failure with PaO2/FiO2 < 300 requiring intubation

Exclusion Criteria:

1. known or high suspicion of pre-existing heart failure, unstable angina
2. presence of severe shock with hemodynamic instability despite escalating vasopressors
3. severe, underlying lung disease (COPD, pulmonary fibrosis, lung cancer. etc.)
4. Concurrent treatments are delivered directly into the lung (ie anesthetics etc)
5. Diagnosis of pulmonary hemorrhage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-11-23 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-10-06 (Actual)

PRIMARY OUTCOMES:
Adverse events (patient) - Decrease in oxygenation | 3 days post-randomization
  Count of any decreases in oxygenation, expressed as PaO2 (mmHg) / FiO2 (% oxygen as a decimal), of greater than 20% during the BLES treatment and up to 30 minutes post-treatment. Change will be calculated relative to pre-treatment values.
Adverse events (patient) - Decrease in hemodynamics | 3 days post-randomization
  Count of any decrease in mean arterial blood pressure >10 mmHg or requirement for >20% increase in vasopressor dose during the BLES procedure and up to 30 minutes post-treatment. Change will be calculated relative to the pre-treatment values.
Adverse event (healthcare worker) - Circuit breach | 3 days post-randomization
  Number of circuit breaches. Count of any circuit breach immediately prior to and during each BLES treatment procedure will be recorded.
Adverse event (healthcare worker) - COVID-19 symptoms | 2 weeks post-randomization
  Count of healthcare personnel involved in the BLES procedure developing symptoms and testing positive for COVID-19.

SECONDARY OUTCOMES:
Change in oxygenation | Every 12 hours post-randomization until ICU discharge or death, whichever comes first, an average of 10 days and assessed up to 30 days.
  PaO2 (in mmHg) / FiO2 (percentage oxygen expressed as a decimal) ratios captured from clinical chart
Change in Lung compliance | Every 12 hours post-randomization until ICU discharge or death, whichever comes first, an average of 10 days and assessed up to 30 days.
  Lung compliance captured from the ventilators, expressed in mL/cm H2O.
Ventilated days | From ICU admission until ICU discharge or death, whichever comes first, an average of 10 days and assessed up to 30 days
  The number of days the patient is receiving mechanical ventilation.
Length of ICU stay | From ICU admission until ICU discharge or death, whichever comes first, an average of 10 days and assessed up to 30 days
  The number of days the patient is admitted to the ICU
Length of hospital stay | From hospital admission until hospital discharge or death, whichever comes first, assessed up to 60 days
  The number of days the patient is admitted to the hospital
Mortality | 30 days
  Number of patients who die within 30 days of ICU admission
G-CSF levels (serum inflammatory biomarker) | ICU day 0, 1, 3 and 7 (7 days)
  G-CSF, in pg/mL, from multiplex cytokine arrays
GM-CSF levels (serum inflammatory biomarker) | ICU day 0, 1, 3 and 7 (7 days)
  GM-CSF, in pg/mL, from multiplex cytokine arrays
IFN gamma levels (serum inflammatory biomarker) | ICU day 0, 1, 3 and 7 (7 days)
  IFN gamma, in pg/mL, from multiplex cytokine arrays
IL-1 beta levels (serum inflammatory biomarker) | ICU day 0, 1, 3 and 7 (7 days)
  IL-1 beta, in pg/mL, from multiplex cytokine arrays
IL-4 levels (serum inflammatory biomarker) | ICU day 0, 1, 3 and 7 (7 days)
  IL-4, in pg/mL, from multiplex cytokine arrays
IL-6 levels (serum inflammatory biomarker) | ICU day 0, 1, 3 and 7 (7 days)
  IL-6, in pg/mL, from multiplex cytokine arrays
IL-10 levels (serum inflammatory biomarker) | ICU day 0, 1, 3 and 7 (7 days)
  IL-10, in pg/mL, from multiplex cytokine arrays
I levels (serum inflammatory biomarker) | ICU day 0, 1, 3 and 7 (7 days)
  I, in pg/mL, from multiplex cytokine arrays
MCP-1 levels (serum inflammatory biomarker) | ICU day 0, 1, 3 and 7 (7 days)
  MCP-1, in pg/mL, from multiplex cytokine arrays
TNF alpha levels (serum inflammatory biomarker) | ICU day 0, 1, 3 and 7 (7 days)
  TNF alpha, in pg/mL, from multiplex cytokine arrays

CONTACTS AND LOCATIONS:
Overall Officials: Jim Lewis, MD, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (2):
- Canada (2):
  - London Health Sciences Centre - University Hospital, London, Ontario
  - Victoria Hospital, London, Ontario

IPD SHARING:
Plan to Share IPD: No